CLINICAL TRIAL: NCT06245512
Title: RECHERCHE DE MARQUEURS DIAGNOSTIQUES ET PRONOSTIQUES DE L'ENDOMETRIOSE DANS LE SANG DES REGLES CHEZ LES FEMMES EN AGE DE PROCREER
Brief Title: Diagnostic and Prognostic Markers of Endometriosis in Menstrual Blood
Acronym: MultiMENDo
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C22-75; 2023-A01857-38 (Other: IDRCB)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis
Keywords: biomarker; diagnosis; prognosis
MeSH Terms: conditions — Endometriosis; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Menstrual blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- With endometriosis: Women affected by endometriosis
- Without endometriosis: Women without any clinical sign of endometriosis

SUMMARY:
The goal of this observational study is to identify diagnostic and prognostic biomarkers for endometriosis using menstrual blood, an easily accessible yet overlooked biological fluid in women of reproductive age, affected or not by endometriosis

The main questions it aims to answer are:

* are there relevant differences in the menstrual blood of women affected by endometriosis compared to women without endometriosis?
* do some of these differences disappear or lessen when the disease is treated by surgery? Participants will answer questions relevant to endometriosis and provide menstrual blood 1 to 3 times (self-collected with a menstrual cup). A subgroup of participants affected by endometriosis that will undergo surgery for their regular care will provide menstrual blood before and after their surgery.

Researchers will compare the menstrual blood of women with and without endometriosis, and before and after surgery to see if they can identify significant differences.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

Women 18-45 of age who

* Have their period
* Have given their written consent
* Have already used a menstrual cup as a method of hygienic protection
* Residing or working in Ile de France (Paris Metropolitan area, France)

For participants with endometriosis:

* diagnosis of endometriosis established by surgery or imaging (ultrasound and/or MRI)
* presence of one or more painful symptoms > 3 on a visual scale (dysmenorrhea and/or dyspareunia and/or chronic pelvic pain) and/or infertility
* for the surgery subgroup: planned surgery in the next 3 months

For participants without endometriosis:

* painful symptoms < or equal to 3 on a visual scale (for dysmenorrhea and dyspareunia and chronic pelvic pain),
* absence of intense period pain in adolescence (leading to taking pills to control this pain and/or peri-menstrual school absenteeism)

Exclusion Criteria:

For all participants:

* Autoimmune diseases
* Chronic diseases other than endometriosis (diabetes, hypertension)
* A person who is the subject of a judicial safeguard measure (by declaration)
* Infectious diseases (HIV, HBV, if known)
* History of menstrual toxic shock syndrome

For patients with endometriosis:

* endometriosis surgery within the last 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women 18-45 of age with periods
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic and prognostic score | 3 years and 8 months
  Score based on candidate biomarkers that will be selected for their quantitative differences between patients with or without endometriosis and for their prognostic potential in the context of response to surgical treatment (significant quantitative difference between before and after surgery). Biomarkers that are both significantly quantitatively different between women with and without endometriosis and before versus after surgery will constitute the final set and this set will be measured by targeted approach in all the participants. This score, associated or not with clinical characteristics (such as for example the intensity of pain, the association of different types of pain), will make it possible to differentiate women with and without endometriosis with a specificity greater than or equal to 79% and a sensitivity greater than or equal to 94%.

SECONDARY OUTCOMES:
Diagnostic score | 3 years and 8 months
  Score based on candidate biomarkers that will be selected for their quantitative differences between patients with or without endometriosis.
Prognostic candidate score | 3 years and 8 months
  Score based on candidate biomarkers that will be selected for their significant quantitative differences between before and after surgery. This score will have to be validated in a bigger cohort in a subsequent clinical study to assess its specificity and sensitivity to differentiate women for who the surgery is effective from women for who the surgery is not or only partially effective, or women with a recurrence of the disease.
Diagnostic score for a specific subtype of endometriosis | 3 years and 8 months
  Score based on candidate biomarkers that will be selected for their quantitative differences between the patients with different subtypes of endometriosis. This score, associated or not with clinical characteristics (such as for example the intensity of pain, the association of different types of pain), will make it possible to differentiate women with a specific subtype of endometriosis with a specificity greater than or equal to 79% and a sensitivity greater than or equal to 94%.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Marcellin, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hopital Cochin, Paris, France